CLINICAL TRIAL: NCT02986074
Title: CompaRison of Paresthesia Mapping to anatomIc Midline-based burSt Programming Strategies
Acronym: CRISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: St Thomas (Ambiguous); Seacroft Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SJM-CIP-10126
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatomical midline lead first (Experimental): subjects in this group will receive stimulation first using an anatomical midline placed lead and subsequently using a paresthesia mapping placed lead
  Interventions: Device: Anatomical midline lead evaluation first
- Paresthesia mapping lead first (Experimental): subjects in this group will receive stimulation first using a paresthesia mapping placed lead and subsequently using an anatomical midline placed lead
  Interventions: Device: Paresthesia mapping lead evaluation first

INTERVENTIONS:
Device: Paresthesia mapping lead evaluation first — Subjects will evaluate the clinical efficacy of stimulation delivered using the lead implanted using paresthesia mapping in the first part of the SCS trial and using the lead implanted using anatomical midline placement in the second part of the SCS trial
  Arms: Paresthesia mapping lead first
Device: Anatomical midline lead evaluation first — Subjects will evaluate the clinical efficacy of stimulation delivered using the lead implanted using anatomical midline in the first part of the SCS trial and using the lead implanted using paresthesia mapping placement in the second part of the SCS trial
  Arms: Anatomical midline lead first

SUMMARY:
The study will compare therapeutic efficacy of a novel spinal cord stimulation leads implant based on anatomical landmarks with standard surgical implantation technique.

DETAILED DESCRIPTION:
The primary purpose of this study is to compare the therapeutic efficacy of the conventional, paresthesia mapping-based burst spinal cord stimulation (SCS) implantation strategy to a more novel, anatomic midline-based approach that has the potential to streamline the workflow associated with the SCS treatment continuum.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent to participate in the study;
* Subject is 18 years of age or older;
* Subject has failed to respond to at least 6 months of conventional treatment including pharmacological treatment, physical therapy, epidural injections and/or radiofrequency therapy as per NICE Tag 0159;
* FBSS subjects with predominant low back pain;
* Subject has a lower back pain intensity of at least 6.0 out of 10.0 on the VAS at baseline;
* Subject is on stable pain medications with a total opioid equivalent of 120 mgs a day or less for at least 28 days prior to enrolling in this study, and is willing to stay on those medications with no dose adjustments until activation of the permanently implanted SCS device;
* Subject's medical record has been evaluated by the Investigator to ensure that the subject is a good candidate for a neurostimulation system;
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all office visits;
* Female candidates of child-bearing potential agree to commit to the use of an effective method of contraception (including but not limited to sterilization, barrier devices, oral contraceptives, intrauterine devices (IUDs), condoms, rhythm method, or abstinence) for the duration of the study

Exclusion Criteria:

* Subjects with significant scoliosis even if surgically corrected
* Subject is currently participating in a clinical investigation that includes an active treatment arm;
* Subject has been implanted with or participated in a trial period for a neurostimulation system;
* Subject has an infusion pump;
* Subject has evidence of an active disruptive psychological or psychiatric disorder as determined as per standard of care;
* Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease or uncontrolled diabetes mellitus;
* Subject has a current diagnosis of a progressive neurological disease as determined by the Investigator;
* Subject is immunocompromised;
* Subject has an existing medical condition that is likely to require repetitive MRI evaluation in the future (i.e. epilepsy, stroke, multiple sclerosis, acoustic neuroma, tumor);
* Subject has history of cancer requiring active treatment in the last 12 months;
* Subject has an existing medical condition that is likely to require the use of diathermy in the future;
* Subject has documented history of allergic response to titanium or silicone;
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection;
* Female candidates of child bearing potential that are pregnant (confirmed by positive urine/blood pregnancy test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lalit Venkatesan, Ph.D., Study Director — Abbott Medical Devices
Locations (2):
- United Kingdom (2):
  - Seacroft Hospital, Leeds, Yorkshire and the Humber
  - St. Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients were enrolled and screened for eligibility between October 2016 and June 2018 in hospitals in London and Leeds U.K.
Pre-assignment Details: 55 of 60 subjects were randomized. Of those not randomized 3 did not meet inclusion criteria, 1 withdrew consent and 1 was withdrawn by the investigator because his diabetes become uncontrolled increasing the risk associated with SCS implant
Groups:
- Anatomical Positioning Lead First: subjects in this group will receive stimulation first using an anatomical midline placed lead and subsequently using a paresthesia mapping placed lead
  Anatomical midline lead evaluation first: Subjects will evaluate the clinical efficacy of stimulation delivered using the lead implanted using anatomical midline in the first part of the SCS trial and using the lead implanted using paresthesia mapping placement in the second part of the SCS trial
- Follow up Using Paresthesia Mapping Lead Stimulation: Subjects that were successful at SCS trial, expressed preference for stimulation delivered using the lead implanted with the paresthesia mapping approach and received permanent implant, were followed up for 12 months while receiving stimulation delivered using the lead implanted with the paresthesia mapping approach
- Follow up Using Anatomical Placement Lead Stimulation: Subjects that were successful at SCS trial, expressed preference for stimulation delivered using the lead implanted with the anatomical positioning approach and received permanent implant, were followed up for 12 months while receiving stimulation delivered using the lead implanted with the anatomical positioning approach
Period: First Trial Period
Arm/Group | Anatomical Positioning Lead First | Paresthesia Mapping Lead First | Follow up Using Paresthesia Mapping Lead Stimulation | Follow up Using Anatomical Placement Lead Stimulation
Started | 26 | 29 | 0 | 0
Completed | 25 | 29 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Second Trial Period
Arm/Group | Anatomical Positioning Lead First | Paresthesia Mapping Lead First | Follow up Using Paresthesia Mapping Lead Stimulation | Follow up Using Anatomical Placement Lead Stimulation
Started | 25 | 29 | 0 | 0
Completed | 25 | 29 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Follow up Period
Arm/Group | Anatomical Positioning Lead First | Paresthesia Mapping Lead First | Follow up Using Paresthesia Mapping Lead Stimulation | Follow up Using Anatomical Placement Lead Stimulation
Started | 0 | 0 | 21 | 22
3 Month Follow up | 0 | 0 | 21 | 21
6 Month Follow up | 0 | 0 | 21 | 20
Completed | 0 | 0 | 20 | 19
Not Completed | 0 | 0 | 1 | 3
Not completed — system explant | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who were enrolled in the study
Arm/Group | All Subjects
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender was not reported for two subjects
  Participants
    number analyzed (Participants) | 53
    Female | 28
    Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 55

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) for Back Pain at SCS Trial
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: after 2 weeks of SCS trial
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Anatomically Positioned Lead: Stimulation delivered using the anatomical lead
- Paresthesia Mapping Lead: Stimulation delivered using the paresthesia mapping lead
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 54 | 54
units on a scale | 32 (25.9) | 30.5 (25.4)

2. Secondary Outcome: Visual Analog Scale (VAS) for Back Pain at 3 Months
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: 3 months after activation of permanent SCS implant
Population: one in the paresthesia mapping lead group had missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 21 | 20
units on a scale | 28.5 (28.1) | 24.6 (19)

3. Secondary Outcome: Visual Analog Scale (VAS) for Back Pain at 6 Months
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: 6 months after activation of permanent SCS implant
Population: Two subjects had missing data in the paresthesia mapping lead group, one patient had missing data in the anatomically positioned lead group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 19 | 19
units on a scale | 24 (24.5) | 35.2 (23.7)

4. Secondary Outcome: Visual Analog Scale (VAS) for Back Pain at 12 Months
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: 12 months after activation of permanent SCS implant
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 19 | 20
units on a scale | 24 (24.5) | 31.8 (26.4)

5. Secondary Outcome: EQ-5D at SCS Trial
Description: Questionnaire on quality of life using european quality of life - 5 dimension questionnaire (EQ-5D) - (Scale is between 0 and 1 with 0 being worse quality of life and 1 best quality of life)
Time Frame: after 2 weeks of SCS trial
Population: Data missing for one patient in the anatomically positioned lead group and one patient for the paresthesia mapping lead group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 53 | 53
score on a scale | 0.68 (0.17) | 0.65 (0.16)

6. Secondary Outcome: EQ-5D at 3 Month
Description: as for outcome 5
Time Frame: 3 months after activation of permanent SCS implant
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 20 | 19
score on a scale | 0.73 (0.2) | 0.63 (0.22)

7. Secondary Outcome: EQ-5D at 6 Month
Description: as for outcome 5
Time Frame: 6 months after activation of permanent SCS implant
Population: One patient had missing data in the anatomically positioned lead group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 19 | 21
score on a scale | 0.62 (0.27) | 0.64 (0.22)

8. Secondary Outcome: EQ-5D at 12 Month
Description: as for outcome 5
Time Frame: 12 months after activation of permanent SCS implant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 19 | 20
score on a scale | 0.69 (0.22) | 0.67 (0.21)

9. Secondary Outcome: ODI at SCS Trial
Description: questionnaire on disability, Oswestry Disability Index (ODI) - (Scale is between 0 and 100 with 0 being no disability and 100 worst disability)
Time Frame: first SCS trial assessment (up to two weeks after electrodes implantation)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 54 | 54
score on a scale | 40.2 (17.1) | 41.8 (16.5)

10. Secondary Outcome: ODI at 3 Months
Description: as for outcome 9
Time Frame: 3 months after activation of permanent SCS implant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 21 | 21
score on a scale | 33.8 (22.6) | 37.3 (20.5)

11. Secondary Outcome: ODI at 6 Months
Description: as for outcome 9
Time Frame: 6 months after activation of permanent SCS implant
Population: One patient had missing data in the anatomically positioned lead group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 19 | 21
score on a scale | 41.5 (23.5) | 36.9 (20.2)

12. Secondary Outcome: ODI at 12 Months
Description: as for outcome 9
Time Frame: 12 months after activation of permanent SCS implant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 19 | 20
score on a scale | 33.9 (21.5) | 39.4 (20.8)

13. Secondary Outcome: Satisfaction Questionnaire
Description: questionnaire regarding patient satisfaction with the therapy
Time Frame: 3 month follow up
Population: One patient had missing data in the paresthesia mapping lead group
Measure: Count of Participants; unit: Participants
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 21 | 20
Participants
  very dissatisfied | 0 | 0
  dissatisfied | 0 | 0
  neither satisfied or dissatisfied | 4 | 1
  satisfied | 8 | 7
  very satisfied | 9 | 12

14. Secondary Outcome: Satisfaction Questionnaire
Description: questionnaire regarding patient satisfaction with the therapy
Time Frame: 6 month follow up
Population: four patients had missing data in the anatomically positioned lead group
Measure: Count of Participants; unit: Participants
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 17 | 21
Participants
  very dissatisfied | 1 | 0
  dissatisfied | 1 | 2
  neither satisfied nor dissatisfied | 4 | 3
  satisfied | 4 | 5
  very satisfied | 7 | 11

15. Secondary Outcome: Satisfaction Questionnaire
Description: questionnaire regarding patient satisfaction with the therapy
Time Frame: 12 month follow up
Population: One patient had missing data in the anatomically positioned lead group
Measure: Count of Participants; unit: Participants
Arm/Group | Anatomically Positioned Lead | Paresthesia Mapping Lead
Number analyzed (Participants) | 18 | 20
Participants
  very dissatisfied | 0 | 0
  dissatisfied | 1 | 1
  neither satisfied nor dissatisfied | 0 | 2
  satisfied | 9 | 4
  very satisfied | 8 | 13

ADVERSE EVENTS:
Time Frame: Through completion of the study, on average about 1 year
Description: Adverse events in this study were not collected per intervention as there were no primary safety endpoints and no investigational devices used in this study.
Groups:
- Anatomically Positioned Leads and Parasthesia Mapped Leads: All subjects enrolled in the study
Arm/Group | Anatomically Positioned Leads and Parasthesia Mapped Leads
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 6/55
Other Adverse Events (participants affected / at risk) | 5/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anatomically Positioned Leads and Parasthesia Mapped Leads (N=55)
abdominal pain due to gall stones (Gastrointestinal disorders) | 1 (1)
difficulty urination and inability to weight bear on right leg (General disorders) | 1 (1)
right leg numbness (General disorders) | 1 (1)
worsening of pain (General disorders) | 1 (1)
photophobia (General disorders) | 1 (1)
wound exploration (Surgical and medical procedures) | 1 (1)
system explant due to suspicion of infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anatomically Positioned Leads and Parasthesia Mapped Leads (N=55)
IPG pain (General disorders) | 3 (4)
headache (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT02986074/Prot_SAP_000.pdf